CLINICAL TRIAL: NCT02505698
Title: A Data Collection Study for the Evaluation of Real Imaging's Real Imager 8 (RI-8) Developed for Risk Assessment of Breast Cancer
Brief Title: A Data Collection Study for the Evaluation of a Novel Infra-red Breast Imaging System for Risk Assessment
Status: Withdrawn | Type: Observational
Why Stopped: Study initiation at this site fell through
Sponsor: Real Imaging Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 960-CLP-ISR-IR8
Record Dates: First submitted 2015-05-04; First posted 2015-07-22 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: Breast Imaging; Mammography; Anatomical Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Three-dimensional functional Metabolic Imaging (3D MIRA) is a new infrared imaging technology using the Real Imager 8 (RI8) developed by Real Imaging. This technology generates 3D metabolic maps of the breast and based on sophisticated machine learning technology, provides objective risk assessment for the presence of malignant tumor in the breast. The procedure is non-invasive, comfortable and does not involve ionizing radiation. It is based on acquiring infrared images of the breast. Those images are processed and analyzed by computers to provide the objective risk assessment.

The technology is intended to be used as a screening tool for breast cancer and emerges as highly useful in women for whom screening mammography is sub-optimal, such as women with dense breast. 3D MIRA is unaffected by breast density and is therefore ideal for evaluating patients with mammographically dense breasts.

Real Imaging is continuously developing the technology including image acquisition hardware and objective analysis of the imaging biomarkers. To further improve and optimize this novel metabolic imaging technology, Real Imaging will introduce an improved imaging device.

The purpose of this clinical study is to collect more imaging data in order to establish superiority of the newer device over the previous one.

The investigators hypothesize is that the new device will be at least as good as the previous one.

DETAILED DESCRIPTION:
Breast cancer remains a leading cause of cancer death among women, with an estimated 1 million new cases and over 400,000 deaths annually worldwide.

In recent years, however, improvements in survival rate have been attributed to earlier diagnosis by national screening programs and better treatments. Although mammography has been the main screening modality of early detection, its limitations such as difficulty in interpreting mammograms for woman with dense breast, are well recognized and the search for more effective technologies for early detection has been receiving increased attention.

Previous studies showed that US (Ultra Sound) can detect more breast cancers not seen on Mammography, particularly in dense breasts. However, breast US sensitivity is not very high and it is highly operator-dependent.

As opposed to US, Breast MRI is highly sensitive, however, it is not used as a screening tool for the general population. The high cost of MRI, its relatively low speciﬁcity (true negative rate), its being time consuming and its need for intravenous contrast agent make it unsuitable as a breast screening tool for the general population.

In light of these shortcomings, the use of the existing screening modalities described that are based on anatomical imaging will result in some misdiagnosis of cancer, particularly in women with dense breast tissue.There is a real need for a novel breast imaging technology that may outperform the current modalities available for women.

The use of infrared imaging for breast cancer screening is an appealing concept, as it is non-invasive, involves no ionization radiation, requires no breast compression and is not affected by breast density. Infrared imaging in the form of thermography, has been utilized in the past for breasts cancer screening with limited success. Detection of thermal asymmetry between breasts, that can point to cancerous tissue, is laborious and inaccurate when examining temperature coded images. Moreover, small focal thermal variations between the breasts causes frequent misdiagnosis.

Real Imaging developed a new infrared imaging technology called 3D MIRA ,(Three-dimensional functional Metabolic Imaging and Risk Assessment) using medical device, Real Imager 8 (RI8). The MIRA technology generates three-dimensional (3D) infrared (IR) metabolic maps of the breast and developed to enable efficient, automated computer analysis of those metabolic maps.

Metabolic imaging will detect signatures of the cancer's microenvironment (e.g angiogenesis). A breast with malignant tumor behaves differently from a healthy breast. In this regard, the breast tumor has specific signatures on the surface of the breast even if the tumor is deeply embedded inside. Metabolic imaging can overcome the limitations of current mammography screening for women with dense breasts. The infrared signal contains information on both anatomical structures and metabolic processes within the breast.

Based on those infrared signals MIRA technology can provide an objective risk assessment for the presence of malignant tumor. The risk assessment is an index that represents the likelihood that a given image dataset includes a malignant finding. The index scale ranges from -100 (normal) to 100 (abnormal). The risk model is based on training the parameters on a calibration set of clinically known cases.

The Real Imager 8.0 (RI8) is composed of two optical heads, each of which includes infrared camera digital camera and video projector. RI8 offers a non-invasive method for Metabolic Imaging and Risk Assessment (MIRA). The RI8 scan enables the determination of risk for breast cancer malignancy, based on assessment of several metabolic parameters. The device does not provide diagnosis or location of cancer. It will offer the physician a support tool to guide the patient to further imaging workup in order to locate, diagnose and characterize the tumor.

The Imaging process is as follows:

The imager is positioned at a distance of approximately 70 cm from the subject who is seated upright throughout the examination. This position will be maintained throughout the imaging session. An initial period of temperature equilibrium precede the imaging process, during which the patient sits in the dedicated imaging room with room temperature set at 18-22 degrees Celsius. Following the temperature equilibration phase, continuous infrared imaging will be acquired for a period of up to 7 minutes. Two minutes after beginning of infrared recording, a metabolic stress test will be induced by having the patient wear cold gloves (0-5 degrees Celsius), which will be removed after 1 minute. This is performed for the purpose of generating vasoconstriction in the breast vessels. The entire imaging session will last approximately 22 minutes. The procedure is comfortable, non-invasive and does not emit or involves any ionizing radiation.

Real Imaging is continuously developing the technology including image acquisition hardware and objective analysis of the imaging biomarkers. To further improve and optimize this novel metabolic imaging technology, Real Imaging will introduce an improved imaging device.

Improvements over the previous approved prototype device include higher resolution and frequency.

Therefore there is a need to collect more imaging data in order to establish superiority of the newer device over the previous one.

The Imaging data will not be used to assess the clinical health status of the volunteers. Data collected during this study is part of Real Imaging's ongoing research and development efforts aimed to create a more effective screening modality for breast cancer.

In this data collection study, approximately 300 female subjects will be enrolled at The Breast Imaging Unit of the Tel-Aviv Medical Center. MIRA's risk assessment will not be provided to the physician nor the subject.

In order to evaluate MIRA's ability to classify healthy women from those who have breast cancer, the enrollment will include two groups:

1. Screening Group - healthy women with no breast findings in previous screening exams
2. Pre-Biopsy Group - women with suspicious findings on recent Mammography and/or US and/or MRI exams with BI-RADS (Breast Imaging-Reporting and Data System) 4/5/6 who are summoned for biopsy for further workup.

Eligible recruited subjects who have signed an informed consent will undergo MIRA imaging prior to being imaged by any other conventional imaging method and if relevant, prior to undergoing a breast biopsy.

MIRA's data of every individual patient will be used for development purposes. The subject's personal, medical, diagnostic examination information and pathology results will be recorded in CRF (case report form) specially designed for this study. Each subject's clinical information will be followed up in order to validate MIRA's results.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Woman has read, understood and signed the inform consent form
* Age: 30 years and older
* Women who are asymptomatic and are scheduled to undergo routine Mx and/or US screening OR Women summoned for breast biopsy following a suspicious finding in recent screening exam and was graded 4/5/6 on BI-RADS scale

Exclusion Criteria:

* Women who have had a Mx (mammography) and/or US and/or MRI examination performed on the day of the study prior to MIRA scan
* Women who had a lumpectomy surgery preceding the study
* Women who had undergone mastectomy and/or breast reconstruction
* Women who have undergone any type of breast surgery preceding the study
* Women who have had a breast biopsy performed throughout the 10 weeks preceding the study
* Women who have a fever on the day of the MIRA imaging
* Women who are pregnant
* Women who are breast-feeding
* Women with implanted pacemaker/defibrillator, implanted venous access device (portacath) or other implanted devices in the chest area
* Women who are unable to read, understand and execute written informed consent
* Women who are have had chemotherapy and/or radiotherapy throughout the 6 months preceding the study

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women aged 30 years and older, and who regardless of this clinical trial are summoned for routine breast cancer screening exam or breast biopsy due to suspicious finding in recent screening exam.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Sufficient number of cancer case and controls have been imaged | up to 12 months
  As this is a data collection study, end point will be reached when approximately 50 women with breast cancer and 100 healthy women (controls) are imaged by the device and sufficient for the comparison statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Orit Golan, MD, Principal Investigator — The Breast Imagning Unit at Tel Aviv Medical Center
Locations (1):
- The Breast Iamging Unit, Tel Aviv, Israel